CLINICAL TRIAL: NCT00378248
Title: Ullevål PersonalityProject. A Randomized Controlled Trial of Intensive Daytreatment Followed by Outpatient Long-term Combined Treatment Compared With Eclectic Individual Therapy for Patients With Personality Disorders
Brief Title: Ullevål PersonalityProject
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPP
Record Dates: First submitted 2006-09-18; First posted 2006-09-19 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Personality Disorders
Keywords: Personality disorders,; Day treatment,; Group psychotherapy,; Combined psychotherapy,; Outcome,; Attachment pattern
MeSH Terms: conditions — Personality Disorders

ARMS (2):
- Combined psychotherapy (Experimental): 18 weeks day hospital treatment followed by long-term outpatient combined group- and individual psychotherapy
  Interventions: Behavioral: Combined psychotherapy
- Outpatient individual psychotherapy (Active Comparator): Eclectic individual psychotherapy in outpatient private practice
  Interventions: Behavioral: Outpatient individual psychotherapy

INTERVENTIONS:
Behavioral: Combined psychotherapy — 18 weeks day hospital treatment followed by long-term outpatient combined group-and individual psychotherapy
  Other Names: CP
  Arms: Combined psychotherapy
Behavioral: Outpatient individual psychotherapy — Eclectic individual psychotherapy in private practice
  Other Names: OIP
  Arms: Outpatient individual psychotherapy

SUMMARY:
Ullevål PersonalityProject is a ranomized controlled trial of treatment of patients with personality disorder. It's main purpose is to test the effect of a long-term combined treatment program compared with eclectic individual therapy for patients with personality disorders.

The main study hypothesis is that long-term combined treatment is superior to eclectic individual therapy with respect to improvement in personality functioning, psychosocial functioning, symptoms, interpersonal problems, and self destructive behavior for poorly functioning patients with personality disorders.

DETAILED DESCRIPTION:
Ullevål PersonalityProject is a ranomized controlled trial of treatment of patients with personality disorder. It's main purpose is to test the effect of a long-term combined treatment program compared with eclectic individual therapy for poorly functioning patients with personality disorders.

The experiment treatment is guided by written treatment guidelines and comprises:

1. 18 weeks intensive day treatment
2. followed by long-term outpatient combined group psychotherapy and individual therapy for 4 and 2,5 years respectively.

The control treatment comprises:

1. eclectic psychotherapy, here understood as psychotherapy according to the preference and regular practice of the therapist.

120 patients with personality disorders admitted to Department of personality psychiatry, Psychiatric division, Ullevål University Hospital are randomized to either experiment or control condition. The patients are evaluated at baseline and after 8, 18, 36, 72 months. The evaluations comprise a large battery of psychological tests and structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* Patients with personality disorders admitted to Department for personality psychiatry, Psychiatric division, Ullevål University Hospital

Exclusion Criteria:

* Schizotypal personality disorder, antisocial personaliy disorder, current alcohol or drug dependence, developmental disorders (e.g. Asperger), symptoms due to organic conditions, and lack of a permanent residence.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2004-05; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Psychosocial functioning | The outcomes will be assessed after 8, 18, 36, and 72 months:
symptom distress | after 8, 18, 36 and 72 months
self esteem | after 8, 18, 36 and 72 months
interpersonal problems, | after 8, 18, 36 and 72 months
self destructive behavior, | after 8, 18, 36 and 72 months
personality pathology, | after 36 and 72 months
quality of life, | after 8, 18, 36 and 72 months
health care utilization after | after 8, 18, 36 and 72 months

SECONDARY OUTCOMES:
affect consciousness | after 36 months
reflective functioning | after 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Wilberg, M.D.Ph.D., Principal Investigator — Oslo University Hospital
Locations (1):
- Department for personality psychiatry, Psychiatric division, Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Result] Arnevik E, Wilberg T, Urnes O, Johansen M, Monsen JT, Karterud S. Psychotherapy for personality disorders: short-term day hospital psychotherapy versus outpatient individual therapy - a randomized controlled study. Eur Psychiatry. 2009 Mar;24(2):71-8. doi: 10.1016/j.eurpsy.2008.09.004. Epub 2008 Dec 19. PMID 19097870
- [Result] Arnevik E, Wilberg T, Urnes O, Johansen M, Monsen JT, Karterud S. Psychotherapy for personality disorders: 18 months' follow-up of the ulleval personality project. J Pers Disord. 2010 Apr;24(2):188-203. doi: 10.1521/pedi.2010.24.2.188. PMID 20420475
- [Result] Gullestad FS, Wilberg T, Klungsoyr O, Johansen MS, Urnes O, Karterud S. Is treatment in a day hospital step-down program superior to outpatient individual psychotherapy for patients with personality disorders? 36 months follow-up of a randomized clinical trial comparing different treatment modalities. Psychother Res. 2012;22(4):426-41. doi: 10.1080/10503307.2012.662608. Epub 2012 Mar 15. PMID 22417131
- [Result] Gullestad FS, Johansen MS, Hoglend P, Karterud S, Wilberg T. Mentalization as a moderator of treatment effects: findings from a randomized clinical trial for personality disorders. Psychother Res. 2013;23(6):674-89. doi: 10.1080/10503307.2012.684103. Epub 2012 May 21. PMID 22612470
- [Result] Gullestad FS, Wilberg T. Change in reflective functioning during psychotherapy--a single-case study. Psychother Res. 2011 Jan;21(1):97-111. doi: 10.1080/10503307.2010.525759. PMID 21331977
- [Derived] Gibbon S, Khalifa NR, Cheung NH, Vollm BA, McCarthy L. Psychological interventions for antisocial personality disorder. Cochrane Database Syst Rev. 2020 Sep 3;9(9):CD007668. doi: 10.1002/14651858.CD007668.pub3. PMID 32880104
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Derived] Klungsoyr O, Antonsen B, Wilberg T. Contours of a causal feedback mechanism between adaptive personality and psychosocial function in patients with personality disorders: a secondary analysis from a randomized clinical trial. BMC Psychiatry. 2017 Jun 5;17(1):210. doi: 10.1186/s12888-017-1365-4. PMID 28583098
- [Derived] Antonsen BT, Klungsoyr O, Kamps A, Hummelen B, Johansen MS, Pedersen G, Urnes O, Kvarstein EH, Karterud S, Wilberg T. Step-down versus outpatient psychotherapeutic treatment for personality disorders: 6-year follow-up of the Ulleval personality project. BMC Psychiatry. 2014 Apr 23;14:119. doi: 10.1186/1471-244X-14-119. PMID 24758722
- [Derived] Kvarstein EH, Arnevik E, Halsteinli V, Ro FG, Karterud S, Wilberg T. Health service costs and clinical gains of psychotherapy for personality disorders: a randomized controlled trial of day-hospital-based step-down treatment versus outpatient treatment at a specialist practice. BMC Psychiatry. 2013 Nov 22;13:315. doi: 10.1186/1471-244X-13-315. PMID 24268099